CLINICAL TRIAL: NCT05092126
Title: Development & Validation of Preoperative Objective Physiological Evaluation
Acronym: POPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00108789
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Cardiorespiratory Fitness
Keywords: areobic power; cardiopulmonary exercise testing; exercise capacity; functional capacity; physical activity
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: All subjects will be asked to complete the exercise test and the fitness questionnaire
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 6MST VO2 (Active Comparator): Completion of 6MST exercise protocol
  Interventions: Behavioral: Exercise
- DASI VO2 (Active Comparator): Completion of DASI fitness activity questionnaire
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Calculate oxygen consumption

SUMMARY:
This study will compare the measured oxygen consumption (VO2) obtained during sub-maximal exercise testing with the estimated VO2 derived from a non-exercise questionnaire.

DETAILED DESCRIPTION:
All surgical patients presenting at the Preoperative Anesthesia & Surgical Screening (PASS Clinic) will complete the Duke Activity Status Index (DASI) self-reported questionnaire as standard of care. If the DASI score is 34 or greater, the patients will not be considered for the study. If the DASI score is 33 or lower, the patient will be considered as a potential study participant. Eligible study participants will then complete a sub-maximal exercise test (Six Minute Step Test, 6MST) with measured VO2.

The VO2 is an integral part of preoperative assessment of cardiorespiratory fitness (CRF). A low CRF is associated with a higher incidence of post-operative complications and mortality. The study will evaluate the ability to estimate VO2 from exercise-derived measurement with questionnaire-derived estimation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Able to speak English
* Ambulatory [assistive devices ok]
* Preoperative Anesthesia and Surgical Screening (PASS) clinic patient with DASI score <34
* Able to provide informed consent

Exclusion Criteria:

* Acute myocardial infarction (3-5 days)
* Unstable angina
* Severe untreated arterial hypertension at rest (>200 mm Hg systolic, >120 mm Hg diastolic)
* Resting heart rate > 120 bpm
* Room air desaturation at rest on room air <85%
* Inmate of correctional facility (i.e. prisoner)
* Diagnosed history of dementia
* Inability to ambulate independently
* Considered inappropriate to participate by Principal Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Total amount of oxygen consumed per minute | Up to 15 minutes
  Oxygen consumption measured in mL/min

CONTACTS AND LOCATIONS:
Overall Officials: David MacLeod, FRCA, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No